CLINICAL TRIAL: NCT00456677
Title: Evaluation of the Utility of Minocycline as an Anti-Inflammatory Agent in the Treatment of Asthma
Acronym: Mino
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: State University of New York - Downstate Medical Center (Other)
Responsible Party: Principal Investigator, Rauno Joks, Associate Professor of Clinical Medicine, State University of New York - Downstate Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Heikki31
Record Dates: First submitted 2007-04-04; First posted 2007-04-05 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Asthma
Keywords: minocycline; asthma; oral corticosteroids
MeSH Terms: conditions — Asthma; cyclopia sequence | interventions — Minocycline

STUDY DESIGN:
Intervention Model Description: Double blind, placebo-controlled. crossover study
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Minocycline (Experimental): Addition of minocycline 150 mg po twice daily to current asthma treatment regimen.
  Interventions: Drug: minocycline
- Placebos (Placebo Comparator): Addition of placebo capsules po twice daily to current asthma treatment regimen
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: minocycline — addition of antibiotic minocycline as antiinflammatory agent in addition to standard of care regimen.
  Other Names: Minocin
  Arms: Minocycline
Drug: Placebos — Addition of oral placebo capsule in addition to standard of care regimen
  Other Names: oral placebo capsules
  Arms: Placebos

SUMMARY:
Trial of effects of minocycline as "add-on" therapy to adults with asthma with a history of requiring at least one episode of oral steroid therapy to control the disease.

DETAILED DESCRIPTION:
This is a double-blind, placebo-controlled crossover study of adult asthmatics given minocycline 150 mg po BID or placebo as add-on therapy for eight weeks each. Each eight week arm is separated by a four week wash-out. Spirometry is performed at the baseline and end of each arm. Daily symptoms scores, peak flow rates, and oral steroid requirements are recorded. A standardized asthma quality of life symptoms assessment is made every four weeks (AQLQ, Juniper).

ELIGIBILITY:
Inclusion Criteria:

* Adult asthmatics
* History of or current use of oral steroids to control symptoms

Exclusion Criteria:

* Pregnant women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 1996-06; Primary Completion 2007-10-01 (Actual); Study Completion 2007-10-01 (Actual)

PRIMARY OUTCOMES:
Decrease in oral steroid therapy requirements. | 8 weeks

SECONDARY OUTCOMES:
improvement in symptoms scores | 8 weeks
  Asthma Quality of Lifes Scores (AQLQ)
improvement in spriometric parameters | 8 weeks
  improvement in spirometric parameters including FEV1, FVC, FEV1/FVC, FEF25-75
improvement in morning and evening peak flow | 8 weeks
decrease in rescue inhaler usage | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rauno Joks, MD, Principal Investigator — State University of New York - Downstate Medical Center
Locations (1):
- SUNY Downstate Medical Center, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No